CLINICAL TRIAL: NCT01537913
Title: Comparison of the Full Outline of UnResponsiveness (FOUR) Score With Glasgow Coma Scale (GCS) in Children With Non-traumatic Impairment of Consciousness.
Brief Title: FOUR Score in Children With Non-traumatic Impairment of Consciousness
Status: Completed | Type: Observational
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Gurpreet Kochar, Comparison of the Full Outline of Unresponsiveness (FOUR) Score and the Glasgow Coma Scale (GCS) in children with non-traumatic impairment of consciousness, All India Institute of Medical Sciences
Other Study IDs: FOUR_Score
Record Dates: First submitted 2012-02-18; First posted 2012-02-23 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2012-02

CONDITIONS: Impaired Consciousness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Hypothesis: FOUR score is a better predictor of outcome (in hospital mortality and functional outcome at discharge) than GCS in children 5- 18 years age admitted in pediatric ward/ ICU with non-traumatic impaired consciousness.

The assessment of comatose patients is an important part of critical care. The assessment of the level of coma relies on clinical scores. The Glasgow Coma Scale (GCS),remains the most commonly used scoring system for altered state of consciousness. Despite its widespread use, a number of limitations have been identified with GCS like inability to assess verbal score in intubated patients and non-inclusion of vital brainstem functions. The FOUR (Full Outline of UnResponsiveness) score, a coma scale consisting of four components (eye response, motor response, brainstem reflexes, and respiration pattern) was recently proposed by investigators from the Mayo Clinic.keeping in view the limitations of GCS, this study was planned to compare the new FOUR score with GCS as a predictor of mortality and poor functional outcome at hospital discharge.

DETAILED DESCRIPTION:
This prospective observational study was carried out from May 2009 to June 2010 in the Department of Pediatrics, All India Institute of Medical Sciences, New Delhi. This study was approved by institutional ethics committee.

Participants We enrolled children aged 5-18 years who presented with impaired consciousness of less than 7 days duration and were admitted in the pediatric ward or pediatric ICU. Children with traumatic brain injury, known vision/hearing impairment, cerebral palsy, mental retardation, degenerative brain disease; those already on sedatives or neuromuscular blockade and with ongoing seizure or seizure within last 1 hour were excluded from the study.

Sample Size From the previous studies, it is known that ROC of GCS in children for prediction of mortality is 0.7.15 Assuming FOUR score to be better predictor of outcome (area under curve for FOUR score assumed to be 0.8), the sample size calculation was done using MedcalcR version 9.2.0.1. The correlation between both the scores and outcome was assumed to be 0.7. Keeping α-level as 0.05 and β-level as 0.20, the sample size was calculated to be 70.

Assessment Procedure The investigator (GK) was trained with the standardized video examples included in a DVD prepared by the developers of the FOUR score (Wijdicks et al10). After training, the investigator demonstrated the score on 2 patients while being supervised by Pediatric Neurologist. There was periodic training of the investigator every month by reviewing the case examples in DVD and rechecking the score periodically.

Written informed consent was obtained from the parents/ guardians for all patients. All the observations (required for the FOUR score and GCS) and investigations (required for PIM2) are done routinely in the children admitted in Pediatric ward/PICU. No additional investigations or interventions were done primarily for the study. Standardized care based on current guidelines was provided to all the patients.

Rater (GK) was given one page hand-out with written instructions describing both the FOUR score and the GCS. The GCS and the FOUR score applied by the rater within two hours of admission and before starting sedatives or neuromuscular blockade. The rater was primary investigator in all the patients. The sequence of application of the scores was randomized using block randomization with block size of 10 patients.

Severity of illness was assessed by PIM2 score16. For PIM2, the values of various variables at time of admission to Pediatric ward/PICU were recorded. PIM 2-based mortality index was evaluated based on the regression equation as published in the literature.The children with impaired consciousness and reduced mental state were classified as obtunded, stuporous or comatose based on classification given by Taylor et al.17 The etiology was determined based on review of the clinical, laboratory and imaging data by the Pediatric Neurologist.

The patient was followed till discharge/ in-hospital mortality. The functional outcome of the patients was assessed by the Pediatric Overall Performance Category (POPC)18 at the time of PICU discharge or 1 month following admission whichever was earlier. This scale ranges in value from 1 to 6 with a value of 1 indicating normal functioning and a value of 6 indicating brain death. Children were considered to have poor outcomes if they scored 3-6 on the POPC scale, consistent with moderate to severe disability to vegetative state, coma or brain death. The POPC score was obtained through direct questions about the child's ability to perform age-appropriate activities, use of rehabilitative services, and physical disabilities.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-18 years
* Meeting the definition of impaired consciousness52
* Admitted in PICU or pediatric ward
* Duration < 7 days

Exclusion Criteria:

* Traumatic brain injury
* Patients already on sedatives or neuromuscular blockade
* Children with cerebral palsy, severe mental retardation, degenerative brain disease.
* Known vision/Hearing impairment
* Ongoing seizures or seizure within last 1 hour

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged 5-18 years, admitted in PICU or pediatric ward with impaired consciousness of less than 7 days duration
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2009-06; Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
In-hospital Mortality | From admission till discharge/ in-hospital mortality

SECONDARY OUTCOMES:
Pediatric Overall Performance Category scale (POPC) scale | 1 month or discharge whichever is earlier

CONTACTS AND LOCATIONS:
Overall Officials: Gurpreet S Kochar, DM, Principal Investigator — All India Institute of Medical Sciences; Sheffali Gulati, Study Director — All India Institute of Medical Sciences; Rakesh Lodha, Study Chair — All India Institute of Medical Sciences